CLINICAL TRIAL: NCT03974256
Title: Evaluation of a New Strategy for the Preparation of Technetium Radioactive Medicaments Using an Innovative Automaton for Nuclear Medicine Examinations: Impact on the Dosimetry of Operators and on the Quality of Preparations
Brief Title: Preparation of Radiopharmaceuticals by Automaton: Operators Dosimetry
Acronym: AUTOTEC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: PHRIP2018/AUTOTEC-GRIGNON-AS
Record Dates: First submitted 2019-05-29; First posted 2019-06-04 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: Exposure, Radiation
Keywords: Automaton; Dosimetry; Radiopharmaceutical; Technetium-99m

STUDY DESIGN:
Intervention Model Description: Interventional study, multicenter, randomized, cross-over, open, at risk and minimal constraints
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group standard method (No Intervention): Operators work during 4 days with thermoluminescent dosimeters (TLD), according to the conventional manual method of preparation of technetium-99m labelled radioactive medicinal products for diagnostic according with good preparation practices and the recommendations contained in the summary of characteristics
- Group automated method (Experimental): Operators work during 4 days with TLD, according to the automated method of preparation of technetium-99m labelled radioactive medicinal products for diagnostic according with good preparation practices and the recommendations contained in the summary of characteristics
  Interventions: Other: Training in the use of the automaton

INTERVENTIONS:
Other: Training in the use of the automaton — 2 days training on automaton use
  Arms: Group automated method

SUMMARY:
The radiopharmaceuticals manipulation used in nuclear medicine department is a significant source of radiation for operators.

According to Article R. 4451-13 of the Labor Code, the exposure limit for hands and skin (average dose over a surface of 1 cm²) received during twelve consecutive months can't exceed the annual dose limit 500 millisieverts (mSv).

The radiopharmaceuticals manipulation exposes operators to the risk of exceeding this limit, as has been shown in a European study.

At present, there are automatons on the market but only for radiopharmaceutical fluorodeoxyglucose (FDG).

One of the advantages of such an automaton is to reduce irradiation of operators' hands during the radiopharmaceuticals preparation. This reduction can reach 95% according to certain authors and the type of automaton.

This study therefore proposes to evaluate the effect of an original, newly designed automaton on operators' dosimetry and the labelled radiopharmaceuticals' quality.

The hypothesis emitted in this study is that the use of this automaton would allow to reduce drastically operators' hands exposure and probably also to improve the precision of the prepared syringes.

This study will be done in a paired way, require a randomization in cross-over and each of the subjects included will be its own witness.

DETAILED DESCRIPTION:
Currently, radiopharmaceuticals for diagnostic purposes are prepared by operators, Technologist in Medical Electro-Radiology or/and Pharmacy Technicians, manually for radiopharmaceuticals labelled with Technetium-99m (99mTc), or using an automaton for radiopharmaceuticals FDG.

At present, there are automatons on the market but only for radiopharmaceuticals FDG.

However, these automatons are currently only used to split into individual doses radiopharmaceuticals FDG, the labelling radiopharmaceuticals being carried out before delivery in nuclear medicine departments.

The Sysark SAS's company has created and patented, with the collaboration of the Center of Research in Automatic Control of Nancy (CRAN, mixed unite of research 7039 common to the University of Lorraine and the CNRS) an innovative automaton for the preparation of radiopharmaceuticals labelled with 99mTc, used to perform scintigraphy examinations of nuclear medicine department.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age > 18 years)
* Operators: Technologist in Electro-Radiology Medical / Pharmacy Technician
* Operators experienced and autonomous in labelling radiopharmaceuticals with technetium-99m, at least one year
* Operators having agreed to participate in the study, having received complete information on the organization of the research and having signed a free and informed consent
* Operators affiliated to a social security scheme or beneficiary of such a scheme

Exclusion Criteria:

* A woman of childbearing age who doesn't have effective contraception
* Persons referred in Articles L. 1121-5, L 1121-8 of the French Public Health Code:

  * Pregnant woman, parturient or mother who is breastfeeding
  * Chil (not emancipated)
  * Adult subject to a measure of legal protection (guardianship, curators, safeguard of justice)
  * Adult unable to express consent
* Persons deprived of their liberty by a judicial or administrative decision, persons under psychiatric care pursuant to Articles L. 3212-1 and L. 3213-1

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Total radiopharmaceutical activity prepared in mega-becquerel (MBq) | Throughout 4 working days of each methods
  For each of the two methods of preparation
Number of days of handling | Throughout 4 working days of each methods
  For each of the two methods of preparation

SECONDARY OUTCOMES:
Accuracy in terms of activity (MBq) of prepared syringes, expressed as a percentage (%) of the prescribed target value, and compared between the automated device and the conventional manual method | Throughout 4 working days of each methods
  For each of the two methods of preparation
A likert of 4 modalities will be used to evaluate the level of comfort in the automaton by operators (from "Very uncomfortable" to "Very comfortable") | After 4 working days of this method
  During the automated method of preparation
A likert of 4 modalities will be used to evaluate the confidence level in the automaton by operators (from "Not at all confident" to "Totally confident") | After 4 working days of each methods
  During the automated method of preparation
Level of operators' irradiation, measured by the breast dosimeter during the 4 days of preparation (in µSv) and expressed in relation to the total radiopharmaceuticals' activity prepared during the same period (in MBq) | Throughout 4 working days of each methods
  For each of the two methods of preparations

CONTACTS AND LOCATIONS:
Overall Officials: Rachel GRIGNON, Technologist, Principal Investigator — GIE NANCYCLOTEP
Locations (1):
- CHRU Nancy - Brabois, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No